CLINICAL TRIAL: NCT01121302
Title: A Phase I Study of Orally-administered AZD5213 in Healthy Males and Non-fertile Females Including Randomized, Double-blind, Placebo-controlled, Parallel-group Assessment of the Safety, Tolerability & PK of Single Ascending Dose (Part 1) & an Open-label Assessment of Effect of Food on the PK (Part 2)
Brief Title: Study to Investigate Single Ascending Oral Doses of AZD5213 in Healthy Male and Non Fertile Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D3030C00001
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Tolerability
Keywords: AZD5213; Phase 1; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): dose escalating
  Interventions: Drug: AZD5213
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5213 — 0.1 mg, 0.3 mg, 1 mg, 2 mg, 4 mg, 8 mg, 16 mg, 32 mg oral solution, single ascending doses
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
1. The main purpose of this study is to assess the safety and tolerability of AZD5213 after single oral doses.
2. Another purpose of this study is to evaluate the pharmacokinetics (also called PK - how the study drug enters and leaves your body and how your body acts on the study drug) of AZD5213 in your blood and urine.

One group of subjects will be studied to see how food affects the pharmacokinetics (PK) of AZD5213 in the blood and urine. They will receive AZD5213 once after fasting overnight and then return to the clinic to receive AZD5213 after eating a high fat breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Suitable veins for cannulation or repeated venipuncture.
* Male healthy volunteers should be willing to use barrier contraception during sexual intercourse, ie condoms, even if partner is using contraceptive method, from the first day of dosing until 3 months after the last dosing with AZD5213.
* Body weight of ≥50 to ≤100 Kg and Body Mass Index (BMI) ≥18 to ≤30 kg/m2.

Exclusion Criteria:

* History and presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastorintestinal and psychiatric/mental disorders.
* History or presence of gastrointestinal (including irritable bowel disease), hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs. Surgery on gastrointestinal tract.
* History of previous or ongoing psychiatric disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs, physical (including neurological) examinations, clinical laboratory variables, electrocardiograms, telemetry, sleep diary (temporal and qualitative aspects), and the Columbia-Suicide Severity Rating Scale | AE will be collected from admission on Day -1 until follow-up

SECONDARY OUTCOMES:
Part 1 : Investigate single-dose PK and dose proportionality of orally-administered AZD5213 | Frequent timepoints within 48 hours of single dose administration
Part 2 Investigate the potential effect of food on AZD5213 PK after administration of AZD5213 as an oral solution | Frequent timepoints after volunteer consumes a high fat, high calorie breakfast, per FDA guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: D3030C00001 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1312&filename=D3030C00001_Clinical_Study_Report_Synopsis.pdf